CLINICAL TRIAL: NCT02852785
Title: 3D Shoulder Kinematics During Throwing-related Movement Patterns Tasks in Upper Extremity Low-to-moderate/Moderate-to-high Loading Conditions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Porto (Other)
Collaborators: University of Lisbon (Other); Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Nuno Morais, PhD student, Universidade do Porto
Other Study IDs: FADEUP_PhDPT_NunoMorais_std#3
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Asymptomatic volleyball attackers: Asymptomatic volleyball attackers involved in competitive events ≥ 2 years and no signs of postural and movement impairments of the upper body quadrant
  Interventions: Behavioral: PNF D2 for flexion; low-to-moderate loading condition; Behavioral: PNF D2 for flexion; moderate-to-high loading condition; Behavioral: PNF D2 for extension; low-to-moderate loading condition; Behavioral: PNF D2 for extension; moderate-to-high loading condition
- Asymptomatic bilateral overhead athletes: Asymptomatic swimmers involved in competitive events ≥ 2 years and no signs of postural and movement impairments of the upper body quadrant
  Interventions: Behavioral: PNF D2 for flexion; low-to-moderate loading condition; Behavioral: PNF D2 for flexion; moderate-to-high loading condition; Behavioral: PNF D2 for extension; low-to-moderate loading condition; Behavioral: PNF D2 for extension; moderate-to-high loading condition
- Asymptomatic non-athletes: Asymptomatic persons not regularly involved in sports activities or occupational overhead tasks (e.g. construction workers),
  Interventions: Behavioral: PNF D2 for flexion; low-to-moderate loading condition; Behavioral: PNF D2 for flexion; moderate-to-high loading condition; Behavioral: PNF D2 for extension; low-to-moderate loading condition; Behavioral: PNF D2 for extension; moderate-to-high loading condition
- Asympt. athletes / scapula dyskinesis: Asymptomatic volleyball attackers involved in competitive events ≥ 2 years and with clinical evidence of scapula dyskinesis
  Interventions: Behavioral: PNF D2 for flexion; low-to-moderate loading condition; Behavioral: PNF D2 for flexion; moderate-to-high loading condition; Behavioral: PNF D2 for extension; low-to-moderate loading condition; Behavioral: PNF D2 for extension; moderate-to-high loading condition
- Symptom. athletes / scapula dyskinesis: Volleyball attackers involved in competitive events ≥ 2 years and with clinical evidence of scapula dyskinesis and complaints of shoulder pain and disability
  Interventions: Behavioral: PNF D2 for flexion; low-to-moderate loading condition; Behavioral: PNF D2 for flexion; moderate-to-high loading condition; Behavioral: PNF D2 for extension; low-to-moderate loading condition; Behavioral: PNF D2 for extension; moderate-to-high loading condition

INTERVENTIONS:
Behavioral: PNF D2 for flexion; low-to-moderate loading condition — Exposure to upper extremity PNF D2 for flexion during low-to-moderate loading condition
Behavioral: PNF D2 for flexion; moderate-to-high loading condition — Exposure to upper extremity PNF D2 for flexion during moderate-to-high loading condition
Behavioral: PNF D2 for extension; low-to-moderate loading condition — Exposure to upper extremity PNF D2 for extension during low-to-moderate loading condition
Behavioral: PNF D2 for extension; moderate-to-high loading condition — Exposure to upper extremity PNF D2 for extension during moderate-to-high loading condition

SUMMARY:
The main purpose of this study is to characterize and compare the 3D shoulder kinematics bilaterally while performing functional movement patterns tests that hypothetically replicate the 5 main phases of the throwing cycle. The tests are based on diagonal D2 for flexion (early and late cocking of the arm) and D2 for extension (acceleration, deceleration and follow-through of the arm) of the upper extremity of proprioceptive neuromuscular facilitation techniques.

DETAILED DESCRIPTION:
The 3D shoulder kinematics (thorax, scapula and humerus) will be collected in different groups of subjects with specific characteristics. To load the upper extremity during PNF D2 for flexion and extension directions, elastic tubing (Thera-Band) will be used as resistance. Selection of the two resistances will be according to a self-perceived ability of the subjects to consistently move a maximal amount of resistance (color) during PNF D2 flexion and extension tests for 15s and 30s, respectively. Each subject will be permitted to sample various resistances in order to assist in selecting the most appropriate load, with no more than three practice repetitions permitted per each resistance sampled.

To perform the tests, subjects will be sited in a standard chair without armrests, with their feet and lower legs placed on another standard chair, positioned just in front of their chair and the non-testing arm placed across the thoracic wall, to minimize the participation of the legs and trunk to upper extremity performance during testing. Elastic tubing will be anchored to a stable base to perform the diagonals (Thera-Band door anchor accessory or the opposite foot). Five repetitions of each test on both sides will be performed, in two different moments (5-10 minutes apart). A rate of 2 seconds per repetition will be employed during recordings using a metronome. A rest period will be given between trials to avoid fatigue. To perform the tests, subjects will begin/end with their hand on the contralateral hip and end/begin at head height and shoulder width. A marker will be placed in the latter position to standardize the start and end of hand position. The order of the tests (PNF D2 flexion and extension) and side (symptomatic/dominant and asymptomatic/non-dominant) will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* subjects who can perform at least 150 degrees of arm elevation

Exclusion Criteria:

* subjects rating pain ≥8/10
* score 5 on any of the items of the Disabilities of Arm, Shoulder and Hand (DASH)
* pain elicited by provocation maneuvers of the neighboring regions (e.g., cervical spine).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes from sports organizations involved in competitive events with pain and disability in the shoulder region
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Side-to-side differences in 3-dimensional scapular angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular position and displacement of the scapula in the 3 planes of [lateral/medial (upward/downward) rotation, protraction/retraction (internal/external rotation), anterior/posterior tilting] at 4 key events of the simulated throwing motion during the two loading conditions (1, initiation of humeral motion; 2, maximum humeral horizontal abduction relative to the trunk; 3, maximum humeral external rotation; 4, maximum humeral internal rotation)
Side-to-side differences in 3-dimensional humerus angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular position and displacement of the humerus in the 3 planes of (plane of elevation, elevation/depression, axial rotation) at 4 key events of the simulated throwing motion during the two loading conditions (1, initiation of humeral motion; 2, maximum humeral horizontal abduction relative to the trunk; 3, maximum humeral external rotation; 4, maximum humeral internal rotation)
Side-to-side differences in 3-dimensional thoracic angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular position and displacement of the thorax in the 3 planes of [flexion/extension, lateral rotation (inclination), axial rotation] at 4 key events of the simulated throwing motion during the two loading conditions (1, initiation of humeral motion; 2, maximum humeral horizontal abduction relative to the trunk; 3, maximum humeral external rotation; 4, maximum humeral internal rotation)

SECONDARY OUTCOMES:
Borg's Rate of Perceived Exertion scale | Through study completion, an average of 1 year
  Rate of Perceived Exertion (RPE) scale varies from 6 (no exertion) to 20 (very, very hard)
Visual Numeric Rating Scale score (0-10) | Through study completion, an average of 1 year
  A 11-point scale to rate pain intensity

CONTACTS AND LOCATIONS:
Locations (3):
- Portugal (3):
  - Faculdade de Motricidade Humana, Universidade de Lisboa, Oeiras, Cruz-Quebrada
  - Escola Superior de Saúde, Instituto Politécnico de Leiria, Leiria
  - Faculdade de Desporto, Universidade do Porto, Porto